CLINICAL TRIAL: NCT00791726
Title: Place of Fundus-related Microperimetry in Uveitic Macular Edema
Brief Title: Microperimetry in Macular Edema
Status: Completed | Type: Observational
Sponsor: St. Franziskus Hospital (Other)
Responsible Party: Department of Ophthalmology at St Franziskus Hospital
Other Study IDs: 2008-448-f-S
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-03

CONDITIONS: Macular Edema; Uveitis
Keywords: microperimetry; macular edema; uveitis; Retinal sensitivity as measured with fundus related microperimetry
MeSH Terms: conditions — Macular Edema; Uveitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with noninfectious uveitis and macular edema

SUMMARY:
In uveitic patients with fluorescein angiographically proven macular edema, a fundus related microperimetry is performed and results are correlated with foveal thickness as measured with optical coherence tomography (OCT).

ELIGIBILITY:
Inclusion Criteria:

* Patients with noninfectious uveitis, macular edema

Exclusion Criteria:

* Pregnancy, fluorescein allergy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with noninfectious uveitis, macular edema
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-11

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology at St Franziskus Hospital, Münster, Northrhine-Westfalia, Germany

REFERENCES:
- [Derived] Roesel M, Heimes B, Heinz C, Henschel A, Spital G, Heiligenhaus A. Comparison of retinal thickness and fundus-related microperimetry with visual acuity in uveitic macular oedema. Acta Ophthalmol. 2011 Sep;89(6):533-7. doi: 10.1111/j.1755-3768.2009.01750.x. Epub 2009 Dec 9. PMID 20003108
- See also: Related Info — http://www.uveitis-zentrum.de